CLINICAL TRIAL: NCT04983095
Title: Metastasis Directed Stereotactic Body Radiotherapy for Oligo Metastatic Hormone Sensitive Prostate Cancer
Acronym: METRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karin Soderkvist (Other)
Collaborators: University Hospital, Umeå (Other); Karolinska University Hospital (Other); Stockholm South General Hospital (Other); Region Skane (Other); Capio Sankt GÃ¶rans Hospital (Unknown); Region Ã-rebro County (Unknown); Ryhov County Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Karin Soderkvist, Senior Consultant, PhD, Umeå University
Organization: Umeå University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METRO_vers1
Record Dates: First submitted 2021-06-01; First posted 2021-07-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer Metastatic; Radiation Therapy; Positron-Emission Tomography
Keywords: Oligometastatic Prostate Cancer; Hormone Sensitive; Stereotactic Body Radiotherapy
MeSH Terms: interventions — Radiosurgery; Radiotherapy, Image-Guided; Androgen Antagonists; Gonadotropin-Releasing Hormone; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Patients are randomised to control (standard care)1:1 intervention (SBRT+standard care)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): ADT+ARPI to all patients and local RT +/- pelvic fields to de novo patients
  Interventions: Combination Product: androgen deprivation therapy; Radiation: Radiotherapy
- SBRT+Standard of Care (Experimental): SBRT to all PSMA+ lesions in addition to SoC and salvage RT to the prostate bed +/- pelvic fields if recurrent post prostatectomy and PSMA-PET+ in the pelvis
  Interventions: Radiation: stereotactic body radiotherapy; Combination Product: androgen deprivation therapy; Radiation: Radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — 30 Gy in 3 fractions alternatively 40 Gy in 5 fractions delivered with stereotactic radiotherapy-principles
  Other Names: stereotactic ablative radiotherapy; image guided radiotherapy
  Arms: SBRT+Standard of Care
Combination Product: androgen deprivation therapy — Medical castration and next-generation Hormonal Agent along with radiotherapy to the prostate in de novo oligometastatic prostate cancer
  Other Names: gonadotropin releasing hormone-agonist; gonadotropin releasing hormone-antagonist; androgen-receptor pathway inhibitor (ARPI)
Radiation: Radiotherapy — RT to the prostate for de novo patients
  Other Names: external radiotherapy

SUMMARY:
The study is an open label, multi-centre, randomized phase III study. The patients will be randomised in a 1:1 ratio to treatment consisting of

* Arm A: MD-SBRT in addition to standard treatment
* Arm B: Standard treatment

Study population: Patients with hormone sensitive prostate cancer (HSPC) with oligometastatic disease detected by PSMA-PET/DT. This includes patients with de novo oligometastatic HSPC and recurrent HSPC after primary RT or prostatectomy.

Primary endpoint: Failure free survival

Secondary endpoints:

* Predictive value of investigated biomarkers in blood and imaging
* Acute and late toxicity after MD-SBRT
* PROM at 3 months, 1, 3 and 5 years
* Castration resistant prostate cancer, CRPC
* Overall survival
* Differences in outcome between patients by strata

Stratification: To avoid imbalance between treatment arms the minimisation method will be used to achieve balance between de novo oligo-metastatic and oligo-recurrent patients, as well as treatment site.

Safety evaluation: Adverse events and side effects graded according to CTCAE v5.0 will be collected every 6th month. Serious Adverse Events are to be reported within 24 hours throughout the study duration.

Statistical methods: Survival endpoints will be calculated using the Kaplan-Meier method with differences compared using the stratified log-rank test. Randomization time is set as baseline time. Pre-planned subgroup analysis will occur based on pre-specified stratification variables. A Cox multivariable regression model will be used to determine factors predictive of survival. Safety analysis will be performed with Mann-Whitney U-test or Fishers exact test.

Criteria for evaluation: Per protocol (patients that have started study treatment) and Intention to treat (all included patients).

Planned sample size: 118 patients

Analysis plan:

The primary end point will be analysed after pre-specified number of events have occurred. All patients randomised to SBRT will be followed minimum 60 months for toxicity. Safety analysis of acute toxicity will take place after median follow up of 6 months. Safety analysis of late toxicity will be analysed after study closure.

Duration of the study:

Three to five years inclusion. 72 months of follow-up after randomization of the last patient.

DETAILED DESCRIPTION:
Standard of Care (arm A and B): 3 years of ADT with the addition of abiraterone+prednisolone for two years. If the patient is de novo oligo-metastatic, RT to the prostate +/- pelvic fields is considered as standard treatment.

Study intervention (arm A): MD-SBRT to all PSMA-PET/CT positive metastatic target volume(s) with 30 Gy in 3 fractions or 40 Gy in 5 fractions in addition to SoC. For recurrent patients post prostatectomy with PSMA-PET-positive finding at prostate bed +/- regional lymph nodes (without prior local RT) salvage RT +/-pelvic fields with SIB to the PSMA+ GTV is to be delivered (sum of SBRT-targets maximum 3).

Screening procedure:Inclusion/exclusion criteria evaluation including evaluation of feasibility of SBRT to all positive lesions on PSMA-PET/CT performed within approx. 30 days of randomization.

Study specific procedure: Recording/collecting of baseline data including baseline PROM and pre-ADT testosterone and PSA. Standard treatment with ADT administered at randomization to all study patients. Abiraterone is initiated within 8 weeks of study entry. Start of MD-SBRT within approx. 28 days of randomization to patients in arm A. Additional RT as specified in study intervention started within 90 days. Follow up according to protocol, minimum 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate cancer (ICD-O-3 C61)
2. WHO/ECOG performance status 0-1
3. 1-3 skeletal or extra pelvic lymph node metastases detected by PSMA-PET/CT in de novo prostate cancer or PSA-relapse after definitive RT or prostatectomy
4. Willing and able to provide informed consent-

Exclusion Criteria:

1. Castration resistant prostate cancer (progression with castrate levels of testosterone)
2. Any treatment known to affect PSA (including ADT) for prostate cancer within 6 months (exception: ADT started due to oligometastatic disease within 2 weeks of study entry)
3. Patient eligible for other treatment (e.g., early docetaxel) than standard treatment described in the protocol as judged by treating physician
4. Life expectancy <3 years by any reason, including concomitant or previous malignancies
5. Previous radiotherapy or surgery that may interfere with the planned treatment (including intra-prostatic recurrence if previous RT to the prostate)
6. > 3 PSMA-PET/CT positive target lesions (excluding the prostate and regional lymph node metastasis in de novo patients or prostate bed and or regional lymph node metastasis in recurrent patients)
7. PSMA-PET verified metastases other than skeletal or lymph nodes
8. Metastases in base of scull and/or calotte
9. Any target lesions not treatable with image guided RT (IGRT) due to overlap with previous RT fields or exceeded dose constraint to OAR(s) as specified in study protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Failure free survival | Throughout the study duration (72 months of follow up for last patient included.)
  Time from randomisation to progressive disease. Progression is defined as 2 consecutive rises in blood PSA. PSA will be collected every third month and registered in the electronic case report form.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5. | Until 6 months after randomisation
  Side effects according to Common Terminology Criteria for Adverse Events version 5, CTCAE v5 will be collected at baseline, 3 and 6 months after randomisation for all organs at risk within 3 cm from the SBRT-target in the electronic case report form. Adverse events are scored from 0 (none) to 5 (fatal) in the electronic case report form. We will report the number of patients with no reported side effects as well as the number of patients scoring 1, 2, 3, 4 and 5 assessed by CTCAE v5.
Number of participants with treatment-related serious adverse events as assessed by CTCAE v5. | Throughout the study duration (72 months of follow up for last patient included.)
  Side effects grade 4 or higher according to Common Terminology Criteria for Adverse Events version 5, CTCAE v5 will be collected every 6th months after randomisation for all organs at risk within 3 cm from the SBRT-target. Adverse events are scored from 0 (none) to 5 (fatal) are collected in the electronic case report form. We will report the number of patients with no reported side effects as well as the number of patients scoring 1, 2, 3, 4 and 5 assessed by CTCAE v5.
Outcome prediction | Throughout the study duration (72 months of follow up for last patient included.)
  Blood samples will be collected to enable evaluation of circulating biomarkers in relation to patient response to treatment at baseline, 1 and 3 months after randomisation, and at progression. Specifically, plasma will be sampled and circulating tumor cells and platelets will be further isolated. Imaging parameters from the baseline PSMA-PET/CT will also be evaluated in relation to outcome.
Patient reported quality of life assessed by EORTC-QLQ 30 | Throughout the study duration (72 months of follow up for last patient included.)
  Patients will fill out a cross validated self registration questionnaire; European Organistaion for Research and Treatment of Cancer Quality of Life Questionnaire, EORTC QLQ 30, at baseline, 3 months, year 1, 3 and 5. The questionnaire consists of 28 statements that are to be graded from 1 (not at all) to 4 (very well) according to how well they correspond to the patients perception. EORTC QLQ30 also ask for the patient to score their overall sense of 1)health and 2)quality of life on a scale from 1 (very poor) to 7 (excellent).
Overall survival | Throughout the study duration (72 months of follow up for last patient included.)
  Death due to any cause
Castration resistent prostate cancer, CRPC | Throughout the study duration (72 months of follow up for last patient included.)
  2 consecutive rises in blood PSA with castrate levels of testosterone. PSA will be collected every third month and registered in the electronic case report form. Testosterone will be collected if a rise in PSA level is detected.

OTHER OUTCOMES:
outcome according to strata | Throughout the study duration (72 months of follow up for last patient included.)
  all outcomes 1-6 will be analysed by stata; primary or recurrent oligometastatic prostate cancer and study site (for inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Söderkvist, Principal Investigator — Region Västerbotten, Umeå University
Locations (7):
- Sweden (7):
  - Region Skåne, Lund, Lund
  - Capio St Göran Hospital, Stockholm, Region Stockholm
  - Södersjukhuset, Stockholm, Region Stockholm
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Umeå University hospital, Umeå, Umea
  - Ryhovs county hospital, Jönköping
  - Region Örebro Län, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: Yes
SBRT-plans will be shared in detail for all treatment related adverse effects grade>3 according to CTCAE vers 5 in both final and interim analyses.
  Study protocol including Statistical Analysis Plan will be made public through per review scientific publication
Supporting Information: Study Protocol, SAP
Time Frame: Planned publication of study at study start
Access Criteria: Open access publication

REFERENCES:
- See also: Official site for clinical trials by Swedish Regional Cancer Centres in Collaboration — https://cancercentrum.se/samverkan/vara-uppdrag/forskning/cancerstudier-i-sverige/